CLINICAL TRIAL: NCT00006045
Title: Phase III, Randomized, Multicenter Study to Assess the Efficacy and Safety of HuM195 (Recombinant Humanized Anti-CD33 Monoclonal Antibody) in Combination With Standardized Chemotherapy Compared to Standardized Chemotherapy Alone in the Treatment of Patients With Refractory or First-Relapsed Acute Myelogenous Leukemia (AML)
Brief Title: Combination Chemotherapy With or Without Monoclonal Antibody Therapy in Treating Patients With Refractory or Relapsed Acute Myelogenous Leukemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Facet Biotech (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068061; PDL-195-301; MSKCC-00029; UCLA-9910050; NCI-G00-1819
Record Dates: First submitted 2000-07-05; First posted 2004-04-13 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2010-02

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute megakaryoblastic leukemia (M7); secondary acute myeloid leukemia; adult acute monocytic leukemia (M5b); adult acute minimally differentiated myeloid leukemia (M0)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — lintuzumab; Cytarabine; Etoposide; Mitoxantrone

INTERVENTIONS:
Biological: lintuzumab
Drug: cytarabine
Drug: etoposide
Drug: mitoxantrone hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. It is not yet known if chemotherapy is more effective with or without monoclonal antibody therapy for acute myelogenous leukemia.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy with or without monoclonal antibody therapy in treating patients who have refractory or relapsed acute myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy, safety, pharmacokinetics, and immunogenicity of mitoxantrone, etoposide, and cytarabine (MEC) with or without monoclonal antibody HuG1-M195 in patients with refractory or relapsed acute myelogenous leukemia.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by age (under 50 vs 50 and over) and duration of previous complete remission (CR) (0-6 vs 7-12 months). All patients receive induction chemotherapy comprised of cytarabine IV over 2 hours, mitoxantrone IV over a maximum of 20 minutes, and etoposide IV over 1-2 hours on days 1-6. On day 5 of induction, patients are randomized to one of two treatment arms: Arm I: Patients receive day 6 of induction chemotherapy. Patients then receive monoclonal antibody HuG1-M195 (MOAB HuM195) IV over 4 hours on days 6-9 or 7-10. Treatment with MOAB HuM195 repeats every 2 weeks for 2 courses (courses 1 and 2) in the absence of disease progression or unacceptable toxicity. During course 1, MOAB HuM195 begins 30 minutes to 24 hours postchemotherapy. Patients who do not achieve CR by day 70 of induction and show evidence of bone marrow progression (regimen failure (RF)) are taken off study. Patients without RF are assigned to one of two consolidation groups based on response: Group A (CR): Patients receive consolidation chemotherapy comprised of mitoxantrone IV over a maximum of 20 minutes on days 1 and 2, and cytarabine IV over 2 hours and etoposide IV over 1-2 hours on days 1-4. Patients with New York Heart Association class II heart disease preconsolidation receive no mitoxantrone during consolidation. Patients receive MOAB HuM195 IV over 4 hours on days 4-7 or 5-8. Treatment with MOAB HuM195 repeats every 2 weeks for 2 additional courses (courses 3 and 4). During course 3, MOAB HuM195 begins 30 minutes to 24 hours postchemotherapy. Group B (partial remission (PR), hematologic improvement (HI), or stable disease (SD)): Patients receive MOAB HuM195 as in group A but no consolidation chemotherapy. Patients without RF after treatment on group A or B receive maintenance MOAB HuM195 IV over 4 hours on days 1-4. Treatment repeats every month for 8 additional courses (courses 5-12). Arm II: Patients receive day 6 of induction chemotherapy. Patients receive no MOAB HuM195 during the entire study. Patients without RF at day 70 of induction are assigned to one of two consolidation groups based on response: Group C (CR): Patients receive consolidation chemotherapy as in group A. Group D (PR, HI, or SD): Patients receive no further treatment. Patients may be eligible to receive MOAB HuM195 on PDL Study 195-302. Patients are followed every 3 months for 1 year, and then every 6 months thereafter.

PROJECTED ACCRUAL: A maximum of 200 patients (100 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven acute myelogenous leukemia (AML) that may have been primary AML, secondary AML, or preceded by hematologic disorder All FAB subtypes except M3 Must meet one of the following three criteria: First relapse within 1 year after documentation of a previous complete remission (CR) achieved by chemotherapy Refractory to prior chemotherapy comprised of a minimum of 1 induction course, including cytarabine at a minimum of 500 mg/m2 (e.g., 100 mg/m2/day for 5 days) plus an anthracycline No high dose cytarabine (no cumulative dose greater than 3 g/m2) First relapse from a previous CR with subsequent autologous bone marrow transplantation (BMT), only if all of the following criteria are met: First BMT At least 100 days but less than 1 year posttransplantation At least 25% cellularity of the bone marrow Previous BMT included full hematopoietic recovery, defined by all of the following: Hemoglobin at least 10 g/dL (without transfusion) Platelet count at least 100,000/mm3 (without transfusion) Absolute neutrophil count at least 1,500/mm3 No transplantation candidates Bone marrow blasts (leukemic cells) greater than 10% No chronic myelogenous leukemia in blast crisis No active CNS leukemia

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 50-100% Life expectancy: Not specified Hematopoietic: See Disease Characteristics Hepatic: Bilirubin less than 2.0 mg/dL (unless related to Gilbert's disease or due to leukemic infiltration) SGOT or SGPT no greater than 4 times upper limit of normal (unless related to AML) Renal: Creatinine less than 2.0 mg/dL (unless related to AML) Cardiovascular: Left ventricular function normal No unstable cardiac arrhythmias, unstable angina pectoris, or myocardial infarction within the past 6 months No New York Heart Association class III or IV heart disease No electrocardiogram evidence of active ischemia Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 1 month after study HIV negative No other active malignancy requiring therapy No active serious infection that is uncontrolled by antimicrobial therapy Medically stable No significant organ dysfunction

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics At least 30 days since prior experimental biologic therapy (e.g., interleukin-2) No concurrent biologic therapy, including bone marrow transplantation Chemotherapy: See Disease Characteristics For first relapse AML with recent or prior chemotherapy: Prior hydroxyurea given as a short course (up to 48 hours) allowed, if needed, to reduce the peripheral leukocyte count Hydroxyurea must be discontinued prior to study For refractory AML with recent or prior chemotherapy: Greater than 2 weeks since prior chemotherapy except hydroxyurea given as above No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No concurrent radiotherapy Surgery: Not specified Other: No other concurrent experimental therapy Concurrent therapy for other preexisting diseases allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-03

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Levitt, MD, PhD, Study Chair — Facet Biotech
Locations (59):
- United States (40):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - St. Joseph Hospital - Orange, Orange, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Sidney Kimmel Cancer Center, San Diego, California
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Emory Clinic, Atlanta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Louisiana State University School of Medicine, Shreveport, Louisiana
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - North Mississippi Hematology and Oncology Associates, Ltd., Tupelo, Mississippi
  - Washington University Barnard Cancer Center, St Louis, Missouri
  - Nevada Cancer Center, Las Vegas, Nevada
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - West Clinic, P.C., Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (3):
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - Institut Jules Bordet, Brussels
  - U.Z. Gasthuisberg, Leuven
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Health Sciences Centre, Winnipeg, Manitoba
  - Queen Elizabeth II Health Science Center, Halifax, Nova Scotia
  - Princess Margaret Hospital, Toronto, Ontario
- France (2):
  - Centre Hospitalier Regional et Universitaire d'Angers, Angers
  - CHRU de Nancy - Hopitaux de Brabois, Vandœuvre-lès-Nancy
- Germany (5):
  - Universitaetsklinikum Benjamin Franklin, Berlin
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Klinikum Rechts Der Isar/Technische Universitaet Muenchen, Munich
  - Westfaelische Wilhelms-Universitaet, Münster
  - University of Rostock, Rostock
- Academisch Medisch Centrum, Amsterdam, Netherlands
- United Kingdom (4):
  - Addenbrooke's NHS Trust, Cambridge, England
  - Royal Free Hospital, Hampstead, London, England
  - Leeds Teaching Hospital Trust, Leeds, England
  - Christie Hospital N.H.S. Trust, Manchester, England